CLINICAL TRIAL: NCT07111104
Title: Survival Efficacy of Combined Radiotherapy and Immunotherapy in Patients With Metastatic Non-small Cell Lung Carcinoma: an Observational Retrospective Multicenter Study
Brief Title: Survival Efficacy of Combined Radiotherapy and Immunotherapy in Patients With Metastatic Non-small Cell Lung Carcinoma
Acronym: ARIS
Status: Completed | Type: Observational
Sponsor: Hopitaux Prives de Metz, Groupe UNEOS (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-001-UNEOS-Obs
Record Dates: First submitted 2025-07-09; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: non small cell lung cancer; NSCLC; metastatic; radiotherapy; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Immunotherapy; Biological Therapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunotherapy cohort: This group includes patients with metastatic non small cell lung cancer (NSCLC) who received immune checkpoints inhibitors (Nivolumab, Atezolizumab or Pembrolizumab) without any associated radiotherapy during the course of treatment
  Interventions: Drug: Immunotherapy
- Immunotherapy + radiotherapy cohort: This group includes patients with metastatic non-small cell lung cancer (NSCLC) who received immune checkpoint inhibitors (Nivolumab, Atezolizumab, or Pembrolizumab) in combination with radiotherapy. Radiotherapy was delivered either concomitantly or sequentially to immunotherapy.
  Interventions: Drug: Immunotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Immunotherapy — The immunotherapy intervention consists of treatment with immune checkpoint inhibitors, specifically Nivolumab (OPDIVO), Atezolizumab (TECENTRIQ), Pembrolizumab (KEYTRUDA).
  These drugs are monoclonal antibodies that block PD-1 or PD-L1 pathways, aiming to enhance the immune system's ability to recognize and destroy cancer cells. The treatment is administered intravenously according to standard dosing schedules.
  Other Names: Biological Therapy
Radiation: Radiotherapy — The radiotherapy intervention involves targeted delivery of ionizing radiation to metastatic lesions. Radiotherapy may be given either concurrently with immunotherapy or sequentially afterward, depending on the patient's treatment plan. The purpose is to achieve local tumor control and potentially enhance the systemic immune response through immunogenic cell death. Different radiation techniques and dose regimens may be employed based on lesion size, location, and clinical considerations.
  Other Names: Radiation Therapy; External Beam Radiotherapy; Radiation Treatment
  Groups: Immunotherapy + radiotherapy cohort

SUMMARY:
The aim of this retrospective, multicenter, observational study is to evaluate the potential clinical benefit of adding radiotherapy (administered either concomitantly or sequentially) to immunotherapy in patients with metastatic non-small cell lung cancer (NSCLC).

One promising approach involves the integration of radiotherapy into the treatment plan. Radiotherapy is known not only for its cytotoxic local effects, but also for its ability to modulate the tumor microenvironment, increase antigen presentation, and stimulate systemic immune responses.

This study will compare two cohorts of patients with metastatic NSCLC treated in real-world clinical settings. The first cohort includes patients treated with immunotherapy alone, while the second includes those who received immunotherapy in combination with radiotherapy. Radiotherapy may have been administered concurrently or sequentially with respect to immunotherapy, based on clinical judgment.

The primary objective is to determine whether the addition of radiotherapy improves progression-free survival (PFS) by at least 30%, compared to immunotherapy alone. This threshold reflects clinically meaningful differences reported in randomized controlled trials in similar populations and treatment lines. Secondary objectives include overall survival (OS) and exploring predictive factors of treatment response, such as patient demographics, tumor characteristics, mutational status, timing of radiotherapy and abscopal effect evaluation, to refine patient selection for future combination strategies.

Eligible participants are adults with histologically confirmed metastatic NSCLC, treated with first-line or second-line immunotherapy, and with no prior exposure to immunotherapy. Data will be retrospectively collected from medical records, and treatment arms will be assigned based on actual clinical care paths.

Participants will:

* Be retrospectively identified from hospital records.
* Be assigned to one of two cohorts: immunotherapy alone or immunotherapy + radiotherapy (concomitant or sequential).
* Have their data analyzed for OS, PFS, toxicity, and potential predictive biomarkers.

The results of this study will contribute to a better understanding of real-world outcomes in metastatic NSCLC patients and may inform future prospective trials evaluating radiotherapy as a modulator of immunotherapy efficacy.

DETAILED DESCRIPTION:
Metastatic non-small cell lung cancer (NSCLC) remains a highly heterogeneous disease with variable responses to immune checkpoint inhibitors, despite their transformative impact on patient outcomes since 2015. Radiotherapy has emerged as a potential synergistic partner for immunotherapy, based not only on its established local cytotoxic effects but also on its capacity to modulate the tumor microenvironment and activate systemic anti-tumor immunity.

Several preclinical and early clinical studies have illustrated how radiation may increase tumor antigen release, upregulate MHC (Major Histocompatibility Complex) class I molecules, and enhance T-cell priming. The abscopal effect, while rare, underscores the possibility that localized radiotherapy can induce immune-mediated tumor regression at distant, non-irradiated sites. These observations support a growing rationale for combining immune checkpoint inhibitors with radiotherapy in a therapeutic strategy that goes beyond additive effects, aiming instead for immune potentiation.

This retrospective, multicenter, observational study investigates whether real-world integration of radiotherapy into immunotherapy regimens improves survival outcomes in patients with metastatic NSCLC. The study is designed to reflect routine clinical practices across participating institutions, with radiotherapy administration (either concomitant or sequential) guided by multidisciplinary clinical decision-making rather than protocolized intervention. This pragmatic approach allows for exploration of a wide range of clinical scenarios and patient profiles, including variation in timing, dose, target site, and sequence of the radiotherapy-immunotherapy combination.

In addition to comparing overall survival (OS) and progression-free survival (PFS) between patients treated with immunotherapy alone versus those receiving additional radiotherapy, the study also seeks to characterize patterns of treatment response, including tumor control in non-irradiated sites, and to identify subgroups most likely to benefit from the combination strategy. Particular interest lies in the immune effect beyond the radiation field, which could serve as an indirect marker of enhanced systemic immune activation.

This study not only aims to generate meaningful insights into real-world treatment patterns and outcomes but also to provide a foundation for future prospective clinical trials. By better understanding how radiotherapy might modulate the immunotherapeutic response in metastatic NSCLC, we hope to refine patient selection, optimize treatment timing, and ultimately improve the effectiveness of immunotherapy in this challenging clinical setting.

Data will be extracted retrospectively from medical records and institutional databases. Collected data will include:

* Demographics: age, sex, smoking history
* Clinical data: performance status, TNM stage (classification system for classifying malignancy), histology, PD-L1 (Programmed Cell Death Ligang 1) status
* Immunotherapy details: agent, start date, treatment duration
* Radiotherapy details: date, site, dose, technique, concurrent/sequential timing
* Survival endpoints: OS (from start of immunotherapy to death), PFS (from start of immunotherapy to radiologic progression or death)
* Adverse events graded by CTCAE (Commun Terminology Criteria for Adverse Events) criteria
* Imaging reports and tumor response: RECIST v1.1 (Response Evaluation Criteria In Solid Tumor) or iRECIST

Statistical Analyses:

* Descriptive statistics: means, medians, frequencies
* Kaplan-Meier analysis for OS and PFS
* Cox proportional hazards regression for hazard ratio estimates
* Subgroup analyses by timing of radiotherapy, PD-L1 level, and other covariates
* Multivariate analysis adjusting for confounders A propensity score matching technique will be used to minimize selection bias by balancing key baseline characteristics between treatment groups. This will allow a more accurate estimation of the effect of radiotherapy, independent of potential confounders such as PD-L1 expression, histologic subtype, and performance status. Outcomes will be assessed in accordance with standardized criteria, and all imaging will be reviewed in multidisciplinary tumor boards to ensure consistency.

Ethical considerations:

This is a non-interventional study using retrospective, anonymized data. No additional procedures or patient contact are required. Institutional approvals and data protection regulations will be respected at all participating centers. The study complies with the General Data Protection Regulation (GDPR) and French data privacy laws.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient with metastatic non-small cell cancer who has received one line of immunotherapy (PEMBROLIZUMAB, ATEZOLIZUMAB and NIVOLUMAB) in stage IV.
* Disease evaluable according to iRECIST v1.1 criteria
* For previously irradiated patients, a non-irradiated lesion evaluable according to iRECIST
* WHO (World Health Organization) score less than or equal to 2.

Exclusion Criteria:

* Composite cancer, small cell lung cancer
* Not metastatic at the time of immunotherapy
* Has already received one line of immunotherapy for non-small cell lung cancer: antibody against Programmed cell Death protein 1 (anti-PD-1), antibody against Programmed Death-Ligand 1 or 2 (anti-PD-L1 and anti-PD-L2), antiboby against Cluster of Differentiation 137 (anti-CD137), antibody against Cytotoxic T-lymphocyte-antigen-4 (anti-CTLA-4)) .
* Second active cancer under treatment
* Immunotherapy for another cancer
* Withdrawal of consent

Non inclusion Criteria:

- Patients treated with DURVALUMAB, on the basis of its marketing authorisation in non-small cell lung cancer and in the adjuvant treatment of NSCLC treated with concomitant radiochemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic non-small cell lung cancer receiving immunotherapy at the metastatic stage, with no previous immunotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 18 months from start of immunotherapy
  PFS is defined as the time from the first administration of immunotherapy to the date of confirmed disease progression or death from any cause, whichever occurs first. Progression is assessed using imaging (CT scan, PET scan or MRI) according to iRECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall Survivall (OS) | Up to 18 months from start of immunotherapy
  OS is defined as the time from the first administration of immunotherapy to the date of death from any cause.
Objective Response Rate (ORR) | Up to 18 months from start of immunotherapy
  ORR is defined as the best tumor response observed during treatment according to iRECIST v1.1 criteria.
  Responses are evaluated based on routine imaging (CT scan, PET scan or MRI) and classified into 5 categories: complete response (iCR), partial response (iPR), stable disease (iSD), unconfirmed progressive disease (iUPD) and confirmed progressive disease (iCPD).
Objective Response Rate (ORR bis) | Up to 18 months from start of immunotherapy
  ORR bis is defined in patients receiving both immunotherapy and radiotherpy and refers to the evaluation of the abscopal effect, i.e. tumor response in non-irradiated lesions according to iRECIST v1.1 criteria.
  Responses are evaluated based on routine imaging (CT scan, PET scan or MRI) and classified into 5 categories: complete response (iCR), partial response (iPR), stable disease (iSD), unconfirmed progressive disease (iUPD) and confirmed progressive disease (iCPD).
Progression Free Survival 2 (PFS-2) | Up to 18 months from start of immunotherapy
  PFS-2 is defined as the time from the start the therapy following immunotherapy to the date of confirmed disease progressipn or death from any cause, whichever occurs first.
  Progression is assessed using imaging (CT scan, PET scan or MRI) according to iRECIST v1.1 criteria.
Progression Free Survival after Radiotherapy (PFS RT) | Up to 18 months from end of radiotherapy.
  PFS-RT is defined as the time from the end of radiotherapy to the date of confirmed disease progression or death from any cause, whichever occurs first.
  Progression is assessed using imaging (CT scan, PET scan or MRI) according to iRECIST v1.1 criteria.
Frequency and severity of toxicities of combined immunotherapy and radiotherapy, according to CTCAE v5.0 grades | Up to 18 months from start of immunotherapy
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care and activities of daily living (ADL).
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to adverse events (AE).

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Guignard, Resident, Principal Investigator — Hopitaux privés de Metz - UNEOS
Locations (1):
- Hopitaux Privés de Metz - UNEOS, Vantoux, France

IPD SHARING:
Plan to Share IPD: No